CLINICAL TRIAL: NCT04174638
Title: Effect of Motivational Interviewing and Education Based on Watson's Theory of Human Caring in Individuals Receiving Hemodialysis: Randomized Controlled Trial
Brief Title: The Effect of Motivational Interviewing and Education Based on Watson's Theory of Human Caring in Hemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Şefika Tuğba YANGÖZ, Principal Investigator, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Akdeniz University
Record Dates: First submitted 2019-07-21; First posted 2019-11-22 (Actual); Results first posted 2021-02-23 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Renal Disease; Adherence, Treatment; Quality of Life; Satisfaction, Patient
Keywords: Compliance; Motivational Interviewing; Models, Nursing; Nursing; Patient Satisfaction; Quality of Life; Randomized Controlled Trial; Renal Dialysis
MeSH Terms: conditions — Kidney Diseases; Treatment Adherence and Compliance; Patient Satisfaction; Patient Compliance | interventions — Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: This study is a parallel group randomized controlled study
Who Masked: Participant
Masking Description: Single blinding was provided that included inclusion criteria and agreement to participate in the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Intervention Group" (Experimental): The intervention group received 15 minute motivational interviewing based on Watson's Theory of Human Caring once a month for 12 weeks and one session 30 minutes education with educational booklet based on Watson's Theory of Human Caring.
  Interventions: Other: Motivational Interviewing and Education Based on Watson's Theory of Human Caring
- "Control Group" (No Intervention): The control group received routine hemodialysis treatment and nursing care in the hemodialysis unit.

INTERVENTIONS:
Other: Motivational Interviewing and Education Based on Watson's Theory of Human Caring — The intervention group received 15 minute motivational interviewing based on Watson's Theory of Human Caring once a month for 12 weeks and one session 30 minutes education with educational booklet based on Watson's Theory of Human Caring. The intervention performed before the hemodialysis session in a separate room in the hemodialysis unit.
  Arms: "Intervention Group"

SUMMARY:
* Motivational interviewing and education based on Watson's Theory of Human Caring have an effect on increasing adherence to fluid intake in individuals receiving hemodialysis treatment.
* Motivational interviewing and education based on Watson's Theory of Human Caring have an effect on increasing adherence to diet in individuals receiving hemodialysis treatment.
* Motivational interviewing and education based on Watson's Theory of Human Caring have an effect on increasing adherence to drug management in individuals receiving hemodialysis treatment.
* Intervention group who receiving Motivational interviewing and education based on Watson's Theory of Human Caring would satisfied with introduced intervention.
* Motivational interviewing and education based on Watson's Theory of Human Caring have an effect on increasing quality of life in individuals receiving hemodialysis treatment.

DETAILED DESCRIPTION:
The intervention group received 15 minute motivational interviewing based on Watson's Theory of Human Caring once a month for 12 weeks and one session 30 minutes education with educational booklet based on Watson's Theory of Human Caring. The control group received usual care. Adherence to fluid intake, diet and drug management, physical parameters and quality of life was measured at baseline and 12th week. The patient satisfaction was measured in the intervention group at 12th week.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were receive hemodialysis at Hemodialysis Unit of University Hospital in Antalya, Turkey
* Patients who had 1 and above from Diet And Fluid Non-Adherence Questionnaire total score
* Patients who had 0 or 1 score from 1.2. and 6. questions or 3., 4. and 5. questions in the Modified Morisky Scale.
* Patients who receiving Hemodialysis treatment for at least 3 months
* Patients who were over 18 years of age,
* Patients who had orientation of individual, place and time
* Patients who were literate
* Patients who no barriers to written or verbal communication
* Patients who agree to participate in the study

Exclusion Criteria:

* Patients who had psychiatric disease
* Patients who had diagnosis of malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-06-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep ÖZER, PhD, RN, Study Director — Akdeniz University
Locations (1):
- Şefika Tuğba Yangöz, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD will share.
Supporting Information: Study Protocol, SAP
Time Frame: starting 1 months after publication
Access Criteria: all people access.

REFERENCES:
- [Background] Tarverdizade Asl P, Lakdizaji S, Ghahramanian A, Seyedrasooli A, Ghavipanjeh Rezaiy S. Effectiveness of Text Messaging and Face to Face Training on Improving Knowledge and Quality of Life of Patients undergoing Hemodialysis: a Randomized Clinical Trial. J Caring Sci. 2018 Jun 1;7(2):95-100. doi: 10.15171/jcs.2018.015. eCollection 2018 Jun. PMID 29977880
- [Background] Kim K, Kang GW, Woo J. The Quality of Life of Hemodialysis Patients Is Affected Not Only by Medical but also Psychosocial Factors: a Canonical Correlation Study. J Korean Med Sci. 2018 Apr 2;33(14):e111. doi: 10.3346/jkms.2018.33.e111. PMID 29607636
- [Background] Marcus C. Strategies for improving the quality of verbal patient and family education: a review of the literature and creation of the EDUCATE model. Health Psychol Behav Med. 2014 Jan 1;2(1):482-495. doi: 10.1080/21642850.2014.900450. Epub 2014 Apr 28. PMID 25750796
- [Background] Nabolsi MM, Wardam L, Al-Halabi JO. Quality of life, depression, adherence to treatment and illness perception of patients on haemodialysis. Int J Nurs Pract. 2015 Feb;21(1):1-10. doi: 10.1111/ijn.12205. Epub 2013 Oct 11. PMID 24124912
- [Background] Beto JA, Schury KA, Bansal VK. Strategies to promote adherence to nutritional advice in patients with chronic kidney disease: a narrative review and commentary. Int J Nephrol Renovasc Dis. 2016 Feb 2;9:21-33. doi: 10.2147/IJNRD.S76831. eCollection 2016. PMID 26893578
- [Background] Efe D, Kocaoz S. Adherence to diet and fluid restriction of individuals on hemodialysis treatment and affecting factors in Turkey. Jpn J Nurs Sci. 2015 Apr;12(2):113-23. doi: 10.1111/jjns.12055. Epub 2014 Aug 13. PMID 25123654
- See also: he effect of nursing counseling on improving knowledge, adherence to treatment and quality of life of patients undergoing hemodialysis. — https://pdfs.semanticscholar.org/a34d/2315956ebfe14b9143275148444c67cbf394.pdf
- See also: Quality of life in hemodialysis patients and the relationship with mortality, hospitalizations and poor treatment adherence — https://europepmc.org/abstract/med/28001183
- See also: The Effect of Nursing Counseling on Improving Knowledge, Adherence to Treatment and Quality of Life of Patients Undergoing Hemodialysis — https://pdfs.semanticscholar.org/a34d/2315956ebfe14b9143275148444c67cbf394.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This randomized controlled study was conducted between April 2019-2020 with total of 60 patients included 32 intervention and 28 control groups who were receiving hemodialysis treatment in the Hemodialysis Unit of Akdeniz University Hospital.
Pre-assignment Details: 60 individuals were randomized into two groups. There were no individuals who did not continue during the follow-up, and no individuals were excluded from the analysis for any reason
Groups:
- Intervention Group: The intervention group received 15 minute motivational interviewing based on Watson's Theory of Human Caring once a month for 12 weeks and one session 30 minutes education with educational booklet based on Watson's Theory of Human Caring.
- Control Group: The control group was given routine hemodialysis treatment and nursing care in the hemodialysis unit.
Period: Overall Study
Arm/Group | Intervention Group | Control Group
Started | 32 | 28
Completed | 32 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 32 intervention and 28 control group were analyzed.
Groups:
- Intervention Group: The intervention group was given 15 minute motivational interviewing for four month period, one session education at the first motivational interviewing and educational booklet based on Watson Human Care Theory.
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 32 | 28 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.12 (17.23) | 51.39 (18.53) | 54.98 (18.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 13 | 24
  Male | 21 | 15 | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 32 | 28 | 60
The duration of hemodialysis treatment [Count of Participants; unit: Participants] — with the sociodemographic questionnaire
  Participants
    3 months-3 years | 18 | 21 | 39
    4-6 years | 9 | 5 | 14
    7 years and over | 5 | 2 | 7
Hemodialysis Access [Count of Participants; unit: Participants] — with the sociodemographic questionnaire
  Participants
    Catheter | 6 | 11 | 17
    Arteriovenous Fistula | 26 | 17 | 43
    Arteriovenous Greft | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Adherence to Fluid Intake on the Fluid Control in Hemodialysis Patients Scale at Week 12
Description: This scale measure adherence to fluid intake.The scale had 24 items and 3 point likert scale. It was included three sub-dimensions: knowledge, behaviors, and attitudes. The knowledge sub-dimension included 7 items and it's score ranged from 7-21. A high score indicates that individuals have higher levels of knowledge about fluid intake. The behavior sub-dimension included 11 items and it's score ranged from 11-33. A high score indicates that individuals' behavior is positive in adherence to fluid intake. The attitudes sub-dimension included 6 items and it's score ranged from 6-18. A high score indicates that individuals' attitudes is positive in adherence to fluid intake. The Fluid Control in Hemodialysis Patients Scale is evaluated on the total score. The lowest and highest score is between 24 and 72. High score indicates that adherence to fluid intake is high.The scale was developed in Turkey. The change between week 12 score and baseline score was reported.
Time Frame: baseline and 12 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 32 | 28
units on a scale
  Knowledge sub-scale | 1.37 (3.54) | -0.17 (1.44)
  Behaviour sub-scale | 3.31 (4.23) | 0.50 (3.92)
  Attitude sub-scale | 6.46 (1.86) | 2.21 (2.52)
  Total score | 11.15 (5.26) | 2.53 (4.72)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Superiority; p < 0.001, t-test, 2 sided — The threshold for statistical significance was p=0.05. The p value was the value of the total score of the Fluid Control in Hemodialysis Patients Scale

2. Primary Outcome: Change From Baseline in Adherence to Diet on the Scale for Dietary Behaviors in Hemodialysis Patients at Week 12
Description: Scale for Dietary Behaviors in Hemodialysis Patients: This scale evaluate adherence to diet management in hemodialysis patients. The scale had 13 items and 5 point likert scale. The score ranged from 13-65. High score indicates that adherence to diet management is high. The scale was developed in Turkey.The change between week 12 score and baseline score was reported.
Time Frame: Baseline and 12 week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 32 | 28
score on a scale | 7.62 (5.51) | 3.10 (4.99)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Superiority; p < 0.001, t-test, 2 sided — The threshold for statistical significance was p=0.05

3. Primary Outcome: Change From Baseline in Adherence to Drug Management on the Modified Morisky Scale at Week 12
Description: Modified Morisky Scale: This scale evaluate adherence to drug management. It is consist of six items and two sub-dimensions:knowledge and motivation. The lowest and highest score is between 0-3 for each sub-dimension. A score higher than zero each sub-dimension indicates high knowledge and motivation in the adherence to drug management. The change between week 12 score and baseline score was reported
Time Frame: Baseline and 12 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 32 | 28
units on a scale
  Knowledge sub-dimension | 1.00 (0.67) | 0.46 (0.50)
  Motivation sub-dimension | 0.68 (0.47) | 0.71 (0.26)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; It was calculated for detect of difference in mean the knowledge sub-dimension score of Modified Morisky Scale between intervention and control group from baseline to week 12; Test type: Superiority; p < 0.001, t-test, 2 sided — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Intervention Group vs Control Group; It was calculated for detect of difference in mean the motivation sub-dimension score of Modified Morisky Scale between intervention and control group from baseline to week 12; Test type: Superiority; p < 0.001, t-test, 2 sided — The threshold for statistical significance was p=0.05

4. Primary Outcome: Change From Baseline in Adherence to Participation in Dialysis Sessions on the Hemodialysis Session Participation Form at Week 4,8,12
Description: Hemodialysis Session Participation Form: This form was used to evaluated the adherence to participation in dialysis sessions at monthly and it was prepared by the researcher. It consisted of yes and no items. If the participant attended all monthly sessions, yes item was marked, if not, no was marked, and the number of sessions did not attend was noted. It was calculated that the mean of the monthly hemodialysis sessions they did not attend.
  The change between week 4, 8, 12 score and baseline score was reported.
Time Frame: baseline and 4, 8, 12 week
Population: This analysis was not performed because all participants in the intervention and control group attended all monthly sessions.
Arm/Group | "Intervention Group" | "Control Group"
Number analyzed (Participants) | 0 | 0

5. Primary Outcome: The Mean of Satisfaction of the Intervention Group From the Introduced Intervention Based on Theory Using Watson Caritas Patient Score at Week 12
Description: Watson Caritas Patient Score: This questionnaire evaluate the satisfaction with nursing care based on Watson's Theory of Human Caring. It is a likert-type form consist of five items. The score of each item ranged from 1-7. As the mean score from each item approaches 7, it shows that individuals are satisfied with care. This questionnaire will perform only to the intervention group. The mean score of the each item of the questionnaire was reported. The data were not collected for this Outcome Measure from participants in the "Control Group" Arm/Group.
Time Frame: 12 week
Population: This analysis was performed to intervention group. Because this questionnaire evaluate the satisfaction with nursing care based on Watson's Theory of Human Caring. The intervention group received nursing care based on Watson's Theory of Human Caring, the control group received routine nursing care that not based on Watson's Theory of Human Caring or other nursing theories.Data were not collected from participants in the Control Group
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Control Group: The control group received routine hemodialysis treatment and nursing care in the hemodialysis unit
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 32 | 0
units on a scale
  Deliver my care with loving-kindness | 6.40 (0.49) |
  Meet my basic human needs. | 6.43 (0.66) |
  Have helping and trusting relationships with me. | 6.34 (0.70) |
  Create a caring environment that helps me to heal. | 6.25 (0.67) |
  Value my personal beliefs and faith, allowing for | 6.37 (0.65) |

6. Primary Outcome: The Mean of Satisfaction From the Motivational Interviewing Evaluated With Motivational Interview Evaluation Form at Week 12
Description: Motivational Interview Evaluation Form: This form was used to evaluated the satisfaction with motivational interviewing and it was prepared by the researcher. This form consists of a item that includes evaluating the motivational interviewing satisfaction with likert scale and two items that include evaluating the inadequacies of the interviewing with open-ended question. The total mean score ranged from 1-5. As the mean score from first item approaches 5, it shows that individuals are satisfied with motivational interviewing.This form will perform only to the intervention group. The mean of the Motivational Interview Evaluation Form was reported.The data were not collected for this Outcome Measure from participants in the "Control Group" Arm/Group.
Time Frame: 12 week
Population: This analysis was performed to intervention group. Because this form evaluate the satisfaction with motivational interviewing. The intervention group received motivational interviewing, the control group received routine nursing care. Data were not collected from participants in the Control Group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 32 | 0
score on a scale | 4.5 (0.5) |

7. Primary Outcome: Change From Baseline in Quality of Life on the Kidney Disease Quality of Life Instrument 36 Scale at Week 12
Description: Kidney Disease Quality of Life Instrument 36 ıtem:This instrument evaluate quality of life of individuals with chronic kidney disease. The KDQOL-36 consists of 36 items and five sub-dimensions: physical and mental functions, kidney disease burden, symptoms and problems, effects of kidney disease on daily life. The scoring of the each sub-scale ranges from 0 to 100. A higher score in each sub-dimension is an indicator of better health and quality of life. The change between week 12 score and baseline score was reported.
Time Frame: baseline and 12 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 32 | 28
units on a scale
  Physical functions sub-dimension | 3.83 (9.33) | 2.36 (6.82)
  Mental functions sub-dimension | 6.60 (9.52) | 3.50 (7.92)
  Burden of kidney disease sub-dimension | 14.06 (22.33) | 4.68 (9.56)
  Symptoms/problems sub-dimension | 11.45 (9.96) | 10.49 (11.31)
  Effects of kidney disease on daily life sub-dimension | 18.74 (15.30) | 13.72 (8.12)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; It was calculated for detect of difference in mean the physical functions sub-dimension score of Kidney Disease Quality of Life Instrument 36 Scale between intervention and control group from baseline to week 12; Test type: Superiority; p = 0.297, t-test, 2 sided — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Intervention Group vs Control Group; It was calculated for detect of difference in mean the mental functions sub-dimension score of Kidney Disease Quality of Life Instrument 36 Scale between intervention and control group from baseline to week 12; Test type: Superiority; p = 0.742, t-test, 2 sided — The threshold for statistical significance was p=0.05
Statistical Analysis 3: Comparison: Intervention Group vs Control Group; It was calculated for detect of difference in mean the burden of kidney disease sub-dimension score of Kidney Disease Quality of Life Instrument 36 Scale between intervention and control group from baseline to week 12; Test type: Superiority; p = 0.719, t-test, 2 sided — The threshold for statistical significance was p=0.05
Statistical Analysis 4: Comparison: Intervention Group vs Control Group; It was calculated for detect of difference in mean the symptoms/problems sub-dimension score of Kidney Disease Quality of Life Instrument 36 Scale between intervention and control group from baseline to week 12; Test type: Superiority; p = 0.063, t-test, 2 sided — The threshold for statistical significance was p=0.05
Statistical Analysis 5: Comparison: Intervention Group vs Control Group; It was calculated for detect of difference in mean the effects of kidney disease on daily life sub-dimension score of Kidney Disease Quality of Life Instrument 36 Scale between intervention and control group from baseline to week 12; Test type: Superiority; p < 0.001, t-test, 2 sided — The threshold for statistical significance was p=0.05

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Intervention Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/28
Other Adverse Events (participants affected / at risk) | 0/32 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-06): https://cdn.clinicaltrials.gov/large-docs/38/NCT04174638/Prot_SAP_000.pdf